CLINICAL TRIAL: NCT07054684
Title: An Open-Label Biomarker Study of BHV-1400 in IgA Nephropathy
Brief Title: Study of BHV-1400 in IgA Nephropathy
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Biohaven Therapeutics Ltd. (Industry)
Responsible Party: Sponsor
Organization: Biohaven Pharmaceuticals, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BHV1400-102
Record Dates: First submitted 2025-06-27; First posted 2025-07-08 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: IgA Nephropathy
Keywords: IgAN; proteinuria; glomerulonephropathy; chronic kidney disease; kidney disease; CKD; nephritis; urologic disease; glomerulonephritis; Glomerular disease; Iga nephropathy; renal disease
MeSH Terms: conditions — Glomerulonephritis, IGA; Proteinuria; Renal Insufficiency, Chronic; Kidney Diseases; Nephritis; Urologic Diseases; Glomerulonephritis

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- BHV-1400 (Experimental)
  Interventions: Drug: BHV-1400

INTERVENTIONS:
Drug: BHV-1400 — BHV-1400 is delivered subcutaneously (SC)

SUMMARY:
The purpose of this study is to determine if BHV-1400 is a safe and tolerable treatment in participants with IgA Nephropathy (IgAN).

ELIGIBILITY:
Key Inclusion Criteria:

1. Participants must have biopsy-confirmed IgA Nephropathy

Key Exclusion Criteria:

1. Any secondary IgAN
2. Any cause of chronic kidney disease not diagnosed as IgAN or due to non-IgAN cause

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Serious AEs (SAEs), AEs leading to discontinuation, deaths | Baseline to Day 29
  To assess the safety and tolerability of BHV-1400. This objective will be measured by assessing the number of unique subjects with SAEs, moderate or severe AEs, AEs leading to discontinuation or deaths
Number of participants with Grade 3-4 treatment-emergent laboratory abnormalities | Baseline to Day 29
  To assess the safety and tolerability of BHV-1400. This objective will be measured by assessing the number of unique subjects with Grade 3 or 4 treatment-emergent laboratory abnormalities.

CONTACTS AND LOCATIONS:
Locations (11):
- United States (10):
  - Site-001, Farmington, Connecticut
  - Site-003, Miami Lakes, Florida
  - Site-011, Miami Lakes, Florida
  - Site-005, Pembroke Pines, Florida
  - Site-008, Lawrenceville, Georgia
  - Site-009, Hinsdale, Illinois
  - Site-012, Indianapolis, Indiana
  - Site-006, Chesterfield, Missouri
  - Site-002, Dakota Dunes, South Dakota
  - Site-004, Houston, Texas
- Site-007, Leicester, United Kingdom